CLINICAL TRIAL: NCT00814502
Title: Does Zolpidem CR Treatment Change Clinical Outcomes in Elderly Hospitalized Patients With Dementia- A Pilot Study
Brief Title: Zolpidem CR and Hospitalized Patients With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Kaloyan Tanev, MD, Neuropsychiatrist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2008-P-001434/1
Record Dates: First submitted 2008-12-18; First posted 2008-12-25 (Estimated); Results first posted 2017-05-22 (Actual); Last update posted 2017-05-22 (Actual); Status verified 2017-04

CONDITIONS: Dementia; Alzheimer Disease; Dementia, Vascular; Sleep Disorders; Circadian Dysregulation
Keywords: Alzheimer disease; Dementia, vascular; Actigraphy; Circadian dysregulation; Sleep Disorders; Circadian rhythm
MeSH Terms: conditions — Dementia; Alzheimer Disease; Dementia, Vascular; Sleep Wake Disorders; Chronobiology Disorders | interventions — Zolpidem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zolpidem CR (Active Comparator): Subjects randomized to Zolpidem CR
  Interventions: Drug: Zolpidem CR
- Placebo (Placebo Comparator): Subjects randomized to Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zolpidem CR — After a 48-hour period of baseline actigraphy and clinical measurements, study subjects were randomized to take either Zolpidem CR 6.25mg by mouth (1 pink tablet) or Placebo by mouth (also 1 pink tablet) for up to 3 weeks or the end of the subjects' hospital stay.
  Other Names: Ambien CR
  Arms: Zolpidem CR
Drug: Placebo — After a 48-hour period of baseline actigraphy and clinical measurements, study subjects were randomized to take either Zolpidem CR 6.25mg by mouth (1 pink tablet) or Placebo by mouth (also 1 pink tablet) for up to 3 weeks or the end of the subjects' hospital stay.
  Arms: Placebo

SUMMARY:
The purpose of this research study is to compare the effectiveness of Zolpidem CR to that of placebo in improving sleep efficiency in people with dementia admitted to the hospital because of their symptoms. You can participate in this study if you have dementia of the Alzheimer's type or vascular dementia. This study involves placebo; a placebo is a tablet that looks exactly like Zolpidem CR, the study drug, but contains no active study drug. We will use placebos to see if the study results are due to the study drug or due to other reasons. Zolpidem CR is also called Ambien CR and is widely available by prescription. Zolpidem CR is approved by the U.S. Food and Drug Administration (FDA) for the short-term treatment of insomnia (trouble falling or staying asleep).

DETAILED DESCRIPTION:
Sleep patterns normally change with age. Sleep/wake cycles appear to be compromised in people suffering from dementia. Most research involving sleep in dementia has involved community dwelling or nursing home residents. Relatively little is known about the sleep patterns of patients with dementia who develop acute behavioral and psychiatric symptoms and necessitate hospitalization. The relationship between sleep disturbances in these patients and behavioral/psychiatric symptoms is also insufficiently studied. The current study will examine these two sets of data (sleep/wake cycles and clinical symptoms) in a population of elderly subjects with Dementia of the Alzheimer's type (DAT) or vascular dementia (VD) during their hospitalization period. We will compare the sleep outcome measures (primarily sleep efficiency) and clinical outcome measures in subjects treated with Zolpidem CR or Placebo. We will utilize a double-blind, randomized, placebo-controlled design to test our hypothesis that targeting sleep disturbances in hospitalized elderly subjects with DAT or VD leads to improvement in sleep and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age between 60-99 years
* Clinical diagnosis of Dementia of the Alzheimer's type or Vascular Dementia
* Only subjects with Mini Mental Status Examination scores of greater or equal to 10 will be enrolled.

Exclusion Criteria:

1. Subjects who are too agitated to be able to wear the activity monitors;
2. Subjects who are actively suicidal or homicidal or for whom the clinical treatment team considers participation in the study to be unsuitable;
3. Subjects with untreated primary sleep disorders;
4. Subjects who receive hypnotic medications during their participation in the study; Subjects who received hypnotic medications prior to enrollment may participate in the study if they agree to stop receiving hypnotic medications (with their attending physician's approval);
5. Subjects who are receiving over the counter sleep aids;
6. Subjects who can not commit to abstaining from alcohol use while in the study;
7. Subjects with known anaphylactic reaction or angioedema with Zolpidem CR.

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kaloyan S Tanev, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McCleery J, Sharpley AL. Pharmacotherapies for sleep disturbances in dementia. Cochrane Database Syst Rev. 2020 Nov 15;11(11):CD009178. doi: 10.1002/14651858.CD009178.pub4. PMID 33189083

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from among the patients admitted to the Massachusetts General Psychiatric inpatient service, Blake 11. Inclusion criteria included age between 60-99 years and a clinical diagnosis of Alzheimer's dementia and/or vascular dementia using DSM-IV criteria.
Pre-assignment Details: 3 subjects signed informed consent (IC) but were never randomized, and are not included in the table below. One changed his mind prior to randomization; another had untreated sleep apnea, discovered the day after he signed IC; the IC of a third subject was not received from her health care proxy until after her discharge from the hospital.
Groups:
- Zolpidem CR: Subjects randomized to Zolpidem CR
  Zolpidem CR: After a 48-hour period of baseline actigraphy and clinical measurements, study subjects randomized to Zolpidem CR received Zolpidem CR 6.25mg by mouth (1 pink tablet) for up to 3 weeks or the end of the subjects' hospital stay.
- Placebo: Subjects randomized to Placebo
  After a 48-hour period of baseline actigraphy and clinical measurements, study subjects randomized to Placebo received Placebo by mouth (also 1 pink tablet) for up to 3 weeks or the end of the subjects' hospital stay.
Period: Overall Study
Arm/Group | Zolpidem CR | Placebo
Started | 8 | 9
Completed | 7 | 7
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Zolpidem CR: Subjects randomized to Zolpidem CR
  Zolpidem CR: After a 48-hour period of baseline actigraphy and clinical measurements, study subjects will be randomized to take either Zolpidem CR 6.25mg by mouth (1 pink tablet) or Placebo by mouth (also 1 pink tablet) for up to 3 weeks or the end of the subjects' hospital stay.
- Placebo: Subjects randomized to Placebo
  Zolpidem CR placebo: After a 48-hour period of baseline actigraphy and clinical measurements, study subjects will be randomized to take either Zolpidem CR 6.25mg by mouth (1 pink tablet) or Placebo by mouth (also 1 pink tablet) for up to 3 weeks or the end of the subjects' hospital stay.
- Total: Total of all reporting groups
Arm/Group | Zolpidem CR | Placebo | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Customized [Count of Participants; unit: Participants]
  Age > = 60 | 8 | 9 | 17
  Age < 60 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 5 | 9
  Unknown or Not Reported | 4 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 7 | 8 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Sleep Efficiency
Description: Sleep efficiency during the down interval. The down interval signifies the period of time (in minutes) at night when subjects are in bed and trying to sleep. Sleep efficiency is calculated as (100*sleep minutes)/[time interval from sleep onset (as defined by the sleep latency) to sleep offset (the end of the last sleep episode in the Down interval)].
  The time period was different for each patient, it was their duration of hospitalization. The first 48 hours patients were not on the study drug, so the reported least squares mean is an estimate of the mean for the subsequent time period where the patients received different therapies. These means are corrected for differences that might have existed during the first 48 hours. The results would be similar to the results attained from considering the mean during the first 48 hours as a baseline covariate in an Analysis of Covariance, but would be more robust to missing data.
Time Frame: Post-intervention, up to 3 weeks
Measure: Least Squares Mean (Standard Error); unit: percentage of sleep (see above)
Groups:
- Zolpidem CR: Subjects randomized to Zolpidem CR
  Zolpidem CR: After a 48-hour period of baseline actigraphy and clinical measurements, study subjects took Zolpidem CR 6.25mg by mouth (1 pink tablet) for up to 3 weeks or the end of the subjects' hospital stay.
- Placebo: Subjects randomized to Placebo
  After a 48-hour period of baseline actigraphy and clinical measurements, study subjects took Placebo by mouth (also 1 pink tablet) for up to 3 weeks or the end of the subjects' hospital stay.
Arm/Group | Zolpidem CR | Placebo
Number analyzed (Participants) | 8 | 9
percentage of sleep (see above) | 75.93 (3.24) | 75.30 (3.14)

2. Primary Outcome: Sleep Minutes
Description: Total sleep minutes during the down period. The down interval signifies the period of time (in minutes) at night when subjects are in bed and trying to sleep.
  The time period was different for each patient, it was their duration of hospitalization. The first 48 hours patients were not on the study drug, so the reported least squares mean is an estimate of the mean for the subsequent time period where the patients received different therapies. These means are corrected for differences that might have existed during the first 48 hours. The results would be similar to the results attained from considering the mean during the first 48 hours as a baseline covariate in an Analysis of Covariance, but would be more robust to missing data.
Time Frame: post-intervention, up to 3 weeks
Measure: Least Squares Mean (Standard Error); unit: sleep minutes
Arm/Group | Zolpidem CR | Placebo
Number analyzed (Participants) | 8 | 9
sleep minutes | 443.71 (30.11) | 422.49 (29.27)

3. Secondary Outcome: Measures of Aggression, Psychosis, General Clinical Status, Cognitive Measures, Mood Symptoms
Description: Rating Scale for Aggressive Behavior in the Elderly (RAGE, 0-61); higher is worse.
  Disruptive Behavior Rating Scales (DBRS, 0-105); higher is worse.
  Neuropsychiatric Inventory (NPI, 0-144) - measures 12 different domains of neuropsychiatric symptoms such as delusions, hallucinations, anxiety, depression, apathy, etc.; higher is worse.
  Montgomery-Asberg Depression Rating Scale (MADRS, 0-90); higher is worse.
  Mini-mental state examination (MMSE, 0-30); higher is better.
  The time period was different for each patient, it was their duration of hospitalization. The first 48 hours patients were not on the study drug, so the reported least squares mean is an estimate of the mean for the subsequent time period where the patients received different therapies. These means are corrected for differences that might have existed during the first 48 hours. The results would be similar to the results attained from considering the mean during the firs
Time Frame: post-intervention, up to 3 weeks
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Zolpidem CR | Placebo
Number analyzed (Participants) | 8 | 9
units on a scale
  NPI Total Score | 18.00 (5.72) | 18.64 (5.36)
  RAGE Total Score | 1.40 (1.31) | 5.82 (2.07)
  DBRS Total Score | 22.64 (0.56) | 22.47 (0.58)
  MMSE Total Score | 24.45 (2.05) | 21.57 (1.93)
  MADRS Total Score | 22.96 (4.75) | 22.56 (4.80)

ADVERSE EVENTS:
Time Frame: Overall time frame of adverse events collection - 4 years, 2 months. Per subject time frame of adverse events collection - duration of study participation - variable length, up to 21 days.
Description: Adverse events were collected by regular investigator assessment, and by medical inpatient chart review of subjects participating in the study.
Arm/Group | Zolpidem CR | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 3/8 | 2/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zolpidem CR (N=8) | Placebo (N=9)
Dizziness (Nervous system disorders) | 2 | 1 — Dizziness, or unsteadiness
Confusion (Nervous system disorders) | 0 | 2 — Confusion, disorientation
Feeling "foggy" or tired (Nervous system disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Small sample size. We were unable to control for different treatments that our subjects received as inpatients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days